CLINICAL TRIAL: NCT07282600
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of Once Weekly Eloralintide in Adult Participants With Obesity or Overweight, and Type 2 Diabetes
Brief Title: A Study of Eloralintide (LY3841136) in Participants With Obesity or Overweight, and Type 2 Diabetes
Acronym: ENLIGHTEN-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27741; J3R-MC-YDAF (Other: Eli Lilly and Company); 2025-523658-15-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Overweight; Obesity
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Eloralintide Dose 1 (Experimental): Participants will receive eloralintide subcutaneously (SC)
  Interventions: Drug: Eloralintide
- Eloralintide Dose 2 (Experimental): Participants will receive eloralintide SC
  Interventions: Drug: Eloralintide
- Eloralintide Dose 3 (Experimental): Participants will receive eloralintide SC
  Interventions: Drug: Eloralintide
- Eloralintide Dose 4 (Experimental): Participants will receive eloralintide SC
  Interventions: Drug: Eloralintide
- Placebo (Placebo Comparator): Participants will receive placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eloralintide — Administered SC
  Other Names: LY3841136
  Arms: Eloralintide Dose 1; Eloralintide Dose 2; Eloralintide Dose 3; Eloralintide Dose 4
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of eloralintide compared with placebo for body weight reduction in participants with overweight or obesity and type 2 diabetes. Participation in the study will last about 75 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes
* Are on stable treatment for type 2 diabetes for at least 90 days prior to screening
* Have a BMI ≥ 27 kg/m2
* Have a stable body weight (<5% body weight change) for 90 days prior to screening

Exclusion Criteria:

* Have a prior or planned surgical treatment for obesity (liposuction, cryolipolysis, or abdominoplasty allowed if performed >1 year before screening)
* Have a prior or planned endoscopic procedure and/or device-based therapy for obesity (prior device-based therapy acceptable if device removal was more than 6 months prior to screening)
* Have type 1 diabetes
* Have taken any of the following antihyperglycemic medications within 90 days before screening:

  * amylin analogs
  * glucagon-like peptide-1 (GLP-1) receptor agonists
  * glucose-dependent insulinotropic polypeptide/glucagon-like peptide-1 (GIP/GLP) receptor agonists, or
  * insulin
* Have had within 90 days prior to screening:

  * heart attack
  * stroke
  * coronary artery revascularization
  * unstable angina, or
  * hospitalization due to congestive heart failure
* Have a history or diagnosis of New York Heart Association Functional Classification Class IV congestive heart failure
* Have taken medications or alternative remedies intended for weight loss within 90 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1035 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 64

SECONDARY OUTCOMES:
Percent Change from Baseline in Total Body Fat Mass | Baseline, Week 64
Change from Baseline in Waist Circumference | Baseline, Week 64
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 64
Percent Change in Baseline in Triglycerides | Baseline, Week 64
Change from Baseline in Systolic Blood Pressure | Baseline, Week 64
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 64
Percent Change from Baseline in High Sensitivity C-Reactive Protein (hsCRP) | Baseline, Week 64
Percent Change from Baseline in Fasting Insulin | Baseline, Week 64
Change in Medication Use | Baseline through Week 64
Change from Baseline in Estimated Glomerular Filtration Rate (eGFR) | Baseline, Week 64
Change from Baseline in Short Form-36 (SF-36 v2) Score | Baseline, Week 64
Change from Baseline in EQ-5D-5L Score | Baseline, Week 64
Change from Baseline in Control of Eating Questionnaire (CoEQ) Score | Baseline, Week 64
Achievement of Improved Categorical Shift in Patient Global Impression of Severity (PGIS) Physical Function Weight | Baseline, Week 64
Pharmacokinetics (PK): Maximum Concentration at Steady State (Cmax,ss) | Baseline through Week 64
PK: Area Under the Concentration Versus Time Curve for One Dosing Interval at Steady State (AUC(0-ᴛ)ss) | Baseline through Week 64

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (159):
- United States (60):
  - Birmingham Clinical Research, Birmingham, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - Tucson Clinical Research Institute, Tucson, Arizona
  - San Fernando Valley Health Institute, Canoga Park, California
  - AMCR Institute, Escondido, California
  - NorCal Medical Research, Inc, Greenbrae, California
  - Inglewood Clinical, Inglewood, California
  - Ark Clinical Research, Long Beach, California
  - Pacific Clinical Studies, Los Alamitos, California
  - Care Access - Santa Clarita, Santa Clarita, California
  - Encompass Clinical Research, Spring Valley, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Care Access - Aurora, Aurora, Colorado
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Arrow Clinical Trials, Daytona Beach, Florida
  - Care Access - Delray Beach, Delray Beach, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Nature Coast Clinical Research - Inverness, Inverness, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Flourish Research Acquisition, LLC dba Flourish Research - North Miami, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Adult Medicine of Lake County, Inc., Mt. Dora, Florida
  - American Research Centers of Florida, Pembroke Pines, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Winter Park, Florida
  - Teak Research Consults - Dunwoody, Dunwoody, Georgia
  - Teak Research Consults, Lawrenceville, Georgia
  - The Jones Center Clinical Research, Macon, Georgia
  - Pacific Diabetes & Endocrine Center, Honolulu, Hawaii
  - NorthShore University Health System, Skokie, Illinois
  - DM Clinical Research - Indianapolis, Indianapolis, Indiana
  - Clinical Trials Management, LLC d/b/a Flourish Research, Metairie, Louisiana
  - IMA Clinical Research Monroe - Armand, Monroe, Louisiana
  - Centennial Medical Group, Columbia, Maryland
  - Lucida Clinical Trials, New Bedford, Massachusetts
  - Clinical Research Professionals, Chesterfield, Missouri
  - Clinvest Headlands Llc, Springfield, Missouri
  - Hypertension & Nephrology Association, Eatontown, New Jersey
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - NYC Research INC, Long Island City, New York
  - PharmQuest Life Sciences, LLC, Greensboro, North Carolina
  - West Clinical Research, Morehead City, North Carolina
  - Trial Management Associates - Wilmington - Floral Parkway, Wilmington, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Care Access - Lima, Lima, Ohio
  - Summit Headlands, Portland, Oregon
  - Preferred Primary Care Physicians, Preferred Clinical Research-St. Clair, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Accellacare - Mt Pleasant, Mt. Pleasant, South Carolina
  - IMA Clinical Research Austin, Austin, Texas
  - Private Practice - Dr. Osvaldo A. Brusco, Corpus Christi, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Diabetes and Thyroid Center of Ft. Worth, Fort Worth, Texas
  - Juno Research, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Research Your Health, Plano, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - Ogden Clinic - Canyon View, Ogden, Utah
  - Diabetes & Endocrine Treatment Specialists, Sandy City, Utah
- Argentina (11):
  - Stat Research S.A., Buenos Aires
  - Investigaciones Medicas Imoba Srl, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires
  - Asociación de Beneficencia Hospital Sirio Libanés, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Instituto Centenario, CABA
  - Centro Diabetológico Dr. Waitman, Córdoba
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - Fundacion Estudios Clinicos, Rosario
  - Instituto Médico Catamarca IMEC, Rosario
- China (15):
  - Luhe Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Pinggu District Hospital, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - The Second Affiliated Hospital Chongqing Medical University, Chongqing
  - Zhujiang Hospital, Guangzhou
  - The Second People's Hospital of Hefei, Hefei
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi
  - Jiangxi Provincial People's Hospital, Nanchang
  - Nanjing First Hospital, Nanjing
  - Jiangsu Province Official Hospital, Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - Jiading District Central Hospital, Shanghai
  - The Second Hospital of Tianjin Medical University, Tianjin
  - Zigong First People's Hospital, Zigong
- Czechia (4):
  - MUDr. Tomas Edelsberger, Krnov
  - MUDr. Miroslav Koliba s.r.o., Ostrava
  - MUDr. Jana Parkanyiova, Prague
  - Diabet2 s.r.o., diabetologicka a interni ambulance, Prague
- Germany (7):
  - Diabetespraxis Dr. Braun, Berlin
  - Private Practice - Dr. Kai Könemann & Dr. Henrik Könemann, Bünde
  - InnoDiab Forschung Gmbh, Essen
  - Diabetes Zentrum Wilhelmsburg, Hamburg
  - Institut für Diabetesforschung GmbH Münster, Münster
  - Schwerpunktpraxis für Diabetes und Ernährungsmedizin Dr. med. Winfried Keuthage, Münster
  - RED-Institut GmbH, Oldenburg
- India (6):
  - Life Care Hospital and Research Centre, Bangalore
  - Belagavi Institute of Medical Sciences - Belagavi, Belgavi
  - Dr. Ram Manohar Lohia Institute of Medical Sciences, Lucknow
  - All India Institute of Medical Sciences (AIIMS) - Nagpur, Nagpur
  - Lifepoint Multispeciality Hospital, Pune
  - Ashirwad Hospital and Research Centre, Ulhasnagar
- Japan (15):
  - Hayashi Diabetes Internal Medicine Clinic, Chigasaki
  - Tokyo-Eki Center-building Clinic, Chūōku
  - Shonan Takai Clinic, Kamakura
  - Oishi Clinic, Kasuya-gun
  - OHAMA Diabetes Clinic, Kawaguchi
  - Higashijujo Sakai Diabetes Internal Medicine Clinic, Kita-ku
  - Tokuyama Clinic, Mihama-ku,Chiba City
  - Shinkenko clinic, Naha
  - Oyama East Clinic, Oyama
  - Shimokitazawa Tomo Clinic, Setagaya-ku
  - Soka Sugiura Internal Medicine Clinic, Sōka
  - Tsuchiura Medical & Health Care Center, Tsuchiura
  - Tsuchiura Beryl Clinic, Tsuchiura
  - Noritake Clinic, Ushiku
  - Yokohama Minoru Clinic, Yokohama
- Mexico (5):
  - Centro de Investigacion Medica de Occidente, S.C., Guadalajara
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad, Guadalajara
  - Unidad de Investigación Clínica y Atención Médica HEPA S.C., Guadalajara
  - Medical Care and Research SA de CV, Mérida
  - Cardiolink Clin Trials, Monterrey
- Poland (8):
  - Niepubliczny Specjalistyczny Zaklad Opieki Zdrowotnej Osrodek Diabetologiczny Popula Spolka Cywilna, Bialystok
  - Centrum Medyczne NEUROMED, Bydgoszcz
  - Ambulatorium Sp. z o.o., Elblag
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczne DIAB-ENDO-MET, Krakow
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - Ekamed, Lublin
  - NZOZ Przychodnia Specjalistyczna Andrzej Wittek, Henryk Rudzki, Ruda Śląska
  - Samodzielny Publiczny Szpital Kliniczny nr 1 SUM, Zabrze
- Puerto Rico (2):
  - Centro de Endocrinologia y Nutricion, Caguas
  - Dorado Medical Complex, Dorado
- Slovakia (6):
  - Diacrin s.r.o., Bratislava
  - MediVet s.r.o., Malacky
  - B-Medical, s.r.o., Námestovo
  - FUNKYSTUFF s.r.o., Nové Zámky
  - DIA-MED CENTRUM s.r.o., Púchov
  - MEDI-DIA s.r.o., Sabinov
- South Korea (6):
  - Korea University Ansan Hospital, Ansan-si
  - The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si
  - Hanyang University Guri Hospital, Guri-si
  - Chosun University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seongnam
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (9):
  - Hospital Universitario de La Ribera, Alzira
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Complejo Hospitalario Ruber Juan Bravo, Madrid
  - H.R.U Málaga - Hospital Civil, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Centro Médico Compostela, Santiago de Compostela
  - Hospital Universitario Virgen Del Rocio, Seville
  - Vithas Hospital Sevilla, Seville
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Eloralintide (LY3841136) in Participants With Obesity or Overweight, and Type 2 Diabetes (ENLIGHTEN-2) — https://trials.lilly.com/en-US/trial/673735